Title: External Tibia Torsion and Passive Muscle Stiffness of Quadriceps as Two Important

Contributors of Joint Loading during Walking in People with Knee Osteoarthritis

NCT number: NCT03628508

Document date: 27-Jul-2020

## The Hong Kong Polytechnic University Department of Rehabilitation Sciences

## Research Project Informed Consent Form

Project title: The effect of altered muscle stiffness and tibia torsion on joint loading in people with knee osteoarthritis

Investigator(s): Name, highest academic degree, and position of all investigators including student(s) of this project must be provided.

FU Siu Ngor, PhD. Associate Professor. Department of Rehabilitation Sciences, The Hong Kong Polytechnic University

Lai Chris, Wai-Keung, PhD, Assistant Professor. Department of Health technology and Informatics, The Hong Kong Polytechnic University

Huang Chen, PhD student. Department of Rehabilitation Sciences, The Hong Kong Polytechnic University

## Project information:

The overall aim of this project is to determine the role of passive muscle mechanical properties and tibial torsion on knee loading during walking.

You will have 3 assessments.

- (1) You will be positioned in supine lying. Your knee will be passively move from 0° to maximal flexion for 6 times. During each movement, an ultrasound transducer will be used to estimate the stiffness of the 3 superficial heads of the thigh muscle.
- (2) You will be required to walk along a 8-meter walkway for 10 times. Before the walk, 16 reflective balls will be positioned on your lower legs. Your walking pattern will be captured by 8 cameras.
- (3) You will be in standing position while perpendicular biplanar radiographs will be conducted.

The evaluation will be conducted at the Duchess of Kent Children Hospital. The total time will be about 1.5 hours

The evaluation will not cause any pain, tiredness nor radiation on your body. The findings from this project enable better understandings on increased joint loading in subjects with knee osteoarthritis. New strategies can be proposed for reducing joint loading on these individuals.

| Consent: | | | | | |
|---|---|---|---|---|---|
| I, | , have | been explained | the details | of this stu | ıdy. I |
| voluntarily consent to pa | articipate in this stu | ıdy. I understan | d that I can v | withdraw fr | om this |
| study at any time withou | t giving reasons, an | d my withdrawal | will not lead | to any puni | ishment |
| or prejudice against me | . I am aware of | any potential risl | k in joining | this study. | I also |
| understand that my person | onal information wi | ill not be disclose | ed to people v | who are not | related |

| to this study and my name or photograph will not appear this study. | on any publications resulted from |
|---|---|
| I can contact the chief investigator, Dr <u>Amy Fu</u> at telephone <u>27666726</u> for any questions about this study. If I have complaints related to the investigator(s), I can contact Ms Vangie Chung, Secretary of the Departmental Research Committee, at 2766 4329. I know I will be given a signed copy of this consent form. | |
| Signature (subject): | Date: |
| Signature (witness): | Date: |